CLINICAL TRIAL: NCT04328337
Title: Investigating Whether Acute Elevation of Fatty Acid Levels Alters Cerebral Glucose Transport and Metabolism
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-2455; 1R01DK123227-01 (NIH)
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-diabetic, normal weight individuals receiving Intralipid (Experimental): Non-diabetic, normal weight individuals receiving Intralipid. Participants will receive an infusion of Intralipid 20% for 12 hours through an IV (prior to and during scan #2)
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Non-diabetic, normal weight individuals receiving saline (Placebo Comparator): Non-diabetic, normal weight individuals receiving saline. Participants will receive an infusion of normal saline (1:1 randomization) at 30 ml/hr for 12 hours through an IV (prior to and during scan #2
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — Infusion of Intralipid 20%
  Arms: Non-diabetic, normal weight individuals receiving Intralipid
Drug: Placebos — saline 30 ml/hr for 12 hours through an IV
  Arms: Non-diabetic, normal weight individuals receiving saline

SUMMARY:
The goal of this study is to understand the role of brain glucose transport in individuals with obesity and the association with cerebral hypometabolism and these individuals' response to plasma glucose elevations. The main premise is that obesity leads to reduced brain glucose transport and that we can measure this reduction with magnetic resonance spectroscopy (MRS). The secondary premises are that this reduction is driven by elevated non esterified fatty acids which act to turn on specific signaling pathways that regulate brain GLUT1 levels.

DETAILED DESCRIPTION:
There are 2 aims of this study. The intent of aim 1 is to measure the effect of obesity on glucose transport and metabolism in the human brain. This study aim will be conducted in non-diabetic, obese individuals and age- and HbA1c-matched normal weight individuals. A total of 15 non-diabetic - normal weight individuals and 15 obese individuals will be enrolled.

The second aim randomizes 40 non-diabetic, normal weight individuals. The intent of aim 2 is to determine whether acute elevation of NEFA levels in lean, healthy individuals will alter cerebral glucose transport. Eligible participants will be randomized (1:1) to receive either intralipid or normal saline.

The focus of this protocol registration is the randomized portion of the study (aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* HbA1C <6.5%
* Normal weight individuals: BMI 17-25 kg/m^2
* Obese individuals: BMI >30 kg/m^2

Exclusion Criteria:

* Creatinine >1.5mg/dL
* Hematocrit <35% for females and <39% for males
* ALT and AST >2.5X upper limit of normal
* Abnormal TSH
* Abnormal PT/PTT/INR
* Triglycerides >200 mg/dL
* Known hepatic, gastrointestinal, renal, neurologic, psychiatric, cerebrovascular disease
* Uncontrolled hypertension
* Current or past 3 months use of ketogenic diet
* Use of any medications, vitamins, or supplements that can alter cerebral metabolism or lipids
* Smoking
* Current or recent steroid use in last 6 months
* >5% body weight change in last 6 months
* Illicit drug use/alcoholism
* Inability to enter MRI/MRS
* For women: pregnancy, seeking pregnancy, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in brain glucose transport capacity | Through End of Study (Up to 12 hours)
  Measurement of brain glucose transport rates using magnetic resonance spectroscopy (MRS).

CONTACTS AND LOCATIONS:
Overall Officials: Janice Jin Hwang, MD, MHS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Biomedical Research Imaging Center Marsico Hall (UNC), Chapel Hill, North Carolina
  - Clinical and Translational Research Center (CTRC) Burnett-Womack Building (UNC), Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No